CLINICAL TRIAL: NCT04485793
Title: Evaluation of the Effect of a Dietary Supplement on Lipid Pattern and Liver Parameters in Moderately Hypercholesterolemic Subjects: a Double-blind, Placebo-controlled, Randomized, Clinical Trial
Brief Title: Effect of a Dietary Supplement on Lipid Pattern and Liver Parameters in Hypercholesterolemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Claudio Borghi, Professor, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NUT1-BO-2019
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator): Dietary supplement
  Interventions: Dietary Supplement: Dietary supplement
- Placebo comparator (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Dietary supplement — Dietary supplement formulated with 400 mg Bergamot d.e. obtained from different parts of the Citrus Bergamot whole fruit (Citrus bergamia Risso et Poiteau, fructus), specifically from fresh fruits collected from November to February (Brumex TM).
  Oral administration: 1 tablet/day at evening meal
  Arms: Active Comparator
Other: Placebo — Oral administration: 1 tablet/day at evening meal
  Arms: Placebo comparator

SUMMARY:
The joint ESC/EAS guidelines for the management of dyslipidaemias recommend, for patients at low/moderate CV risk with raised LDL-C, a set of measures collectively defined as "lifestyle interventions", with use of drugs only if the LDL-C levels cannot be controlled with such lifestyle interventions. "Lifestyle interventions" also includes food supplements. The reason is the following: a simple "dietary advice" has been shown (Cochrane review and meta-analysis, Rees et al, 2013) to achieve a modest reduction of total-C and LDL-C. The review reports: Dietary advice reduced total serum cholesterol by 0.15 mmol/L (95% CI 0.06 to 0.23) and LDL cholesterol by 0.16 mmol/L (95% CI 0.08 to 0.24) after 3 to 24 months." An average reduction of LDL-C by 0.16 mmol/L (6.2 mg/dL) is definitely insufficient to control the level of LDL-C in those subjects. Therefore, those subjects would lose motivation to keep dieting. In this context, use of supplements would significantly amplify the result of diet.

A significant proportion of ischemic cardiovascular events are believed to be supported by the coexistence of traditional cardiovascular risk factors such as diabetes, hypertension, dyslipidemia, smoking, and others. The aggregation of these factors is accompanied by a significant increase in the risk of cardiovascular events.

Observational studies shown the existence of a relationship between cholesterolemia and coronary heart disease, clearly showing that subjects with even modestly increased total cholesterol values over time develop both fatal and non-fatal vascular events with a higher frequency compared to subjects with similar characteristics, but with lower basal values of cholesterol.

Numerous controlled intervention studies, on the other hand, have shown that there is a close correlation between cholesterol reduction and cardiovascular risk; in fact, reductions in the plasma concentration of total and LDL-C, obtained through lifestyle modification or specific drugs, result in reductions in the incidence of major coronary events. The effectiveness of these interventions has been demonstrated both in subjects in primary prevention and in patients in secondary prevention.

ELIGIBILITY:
Inclusion Criteria:

* Subjects agree to participate in the study and having dated and signed the informed consent form.
* Subjects who have the capability to communicate, to make themselves understood, and to comply with the study's requirements.
* Male or female aged ≥ 18 years and ≤ 70 years old.
* LDL-Cholesterol plasma levels >115 mg/dL and < 190 mg/dL.
* TG<400 mg/dL.
* Subjects who, according to the SCORE charts, have a low or moderate cardiovascular risk (defined as a total cardiovascular risk < 5%) and for whom, according to ESC/EAS guidelines 2012, the intervention strategy does not require a pharmacological lipid-lowering intervention.

Exclusion Criteria:

* Subjects already affected by cardiovascular diseases (secondary prevention) or with estimated 10 years cardiovascular disease risk> 5%;
* Obesity (BMI>30 kg/m2) or diabetes mellitus;
* Assumption of lipid lowering drugs or food supplements, or drugs potentially affecting the lipid metabolism;
* Antihypertensive treatment not stabilized since at least 3 months;
* Anticoagulants therapy
* Uncontrolled hypertension (systolic blood pressure> 190 mmHg or diastolic arterial pressure> 100 mmHg);
* Known current thyroid, gastrointestinal or hepatobiliary diseases;
* Any medical or surgical condition that would limit the patient adhesion to the study protocol;
* Abuse of alcohol or drugs (current or previous);
* History of malignant neoplasia in the 5 years prior to enrolment in the study;
* History or clinical evidence of inflammatory disease such as severe arthritis, systemic lupus erythematosus or chronic inflammatory diseases or current therapy with immunosuppressive agents or long-term glucocorticoids;
* History or clinical evidence of any significant concomitant disease that could compromise the safety of the subject or the possibility of completing the study;
* Known previous intolerance to the tested nutraceutical
* Women in fertile age not using consolidated contraceptive methods
* Pregnancy and Breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
LDL-cholesterolemia absolute reduction from baseline and between groups | 12 weeks
  Absolute reduction of LDL-cholesterolemia after 12 weeks of treatment
LDL-cholesterolemia % reduction from baseline and between groups | 12 weeks
  % reduction of LDL-cholesterolemia after 12 weeks of treatment

SECONDARY OUTCOMES:
Absolute reduction from baseline and between groups in other lipid fractions, apolipoproteins and their ratios | 12 weeks
  Absolute reduction of serum concentrations of total cholesterol, HDL-cholesterol, apolipoprotein B, triglycerides and their ratios after 12 weeks of treatment
% reduction from baseline and between groups in other lipid fractions, apolipoproteins and their ratios | 12 weeks
  % reduction of of serum concentrations of total cholesterol, HDL-cholesterol, apolipoprotein B, triglycerides and their ratios after 12 weeks of treatment
% reduction from baseline and between groups in anthropometric parameters | 12 weeks
  % reduction of body mass index after 12 weeks of treatment
% reduction from baseline and between groups in blood pressure levels | 12 weeks
  % reduction of systolic and diastolic blood pressure after 12 weeks of treatment
Absolute reduction from baseline and between groups in blood pressure levels | 12 weeks
  Absolute reduction of systolic and diastolic blood pressure after 12 weeks of treatment
Absolute reduction from baseline and between groups in anthropometric parameters | 12 weeks
  Absolute reduction of body mass index after 12 weeks of treatment
% reduction from baseline and between groups in creatine phosphokinase (CPK) serum levels | 12 weeks
  % reduction of creatine phosphokinase (CPK) serum levels after 12 weeks of treatment
Absolute reduction from baseline and between groups in creatine phosphokinase (CPK) serum levels | 12 weeks
  Absolute reduction of creatine phosphokinase (CPK) serum levels after 12 weeks of treatment
Absolute reduction from baseline and between groups in liver parameters | 12 weeks
  Absolute reduction of GOT, GPT and gamma-GT after 12 weeks of treatment
% reduction from baseline and between groups in liver parameters | 12 weeks
  % reduction of GOT, GPT and gamma-GT after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Borghi, MD, Principal Investigator — S. Orsola-Malpighi University Hospital
Locations (1):
- University of Bologna, Bologna, BO, Italy

REFERENCES:
- [Result] Pierdomenico M, Cicero AFG, Veronesi M, Fogacci F, Riccioni C, Benassi B. Effect of Citrus bergamia extract on lipid profile: A combined in vitro and human study. Phytother Res. 2023 Sep;37(9):4185-4195. doi: 10.1002/ptr.7897. Epub 2023 Jun 13. PMID 37312672